CLINICAL TRIAL: NCT04841993
Title: Pharmacokinetics and Pharmacological Effects of a Standardized Cannabis Preparation in Healthy Adult Recreational Cannabis Users
Brief Title: Pharmacokinetics and Pharmacological Effects of a Standardized Cannabis Preparation
Acronym: CANNMED
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundació Institut Germans Trias i Pujol (Other); Istituto Superiore di Sanità (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HUGTP/CANNMED/1
Record Dates: First submitted 2021-03-03; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Cannabis Use; Healthy Subjects
Keywords: medical cannabis; pharmacokinetics; acute effects; cannabis decoction; cannabis oil; vaporized cannabis; oral cannabis
MeSH Terms: interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: The study was unicentric, open-label, not randomized, not placebo controlled ,single blind. The study included three substudies (one for each formulation administration). The first one for decoction administration, the second one for oil administration, and finally, an experimental session was held for the administration of the standardized vaporized cannabis preparation. Each subject will participate in one experimental session. One treatment condition per subject (of two possible oral formulations and one inhaled / vaporized formulation of vaporized cannabis. Once the experimental session is over, the subjects have the possibility of being able to participate in the same study after a minimum washout period of 3 weeks.
Who Masked: Participant
Masking Description: Participant were aware of the cannabis preparation but not of the administered doses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral formulation: Cannabis decoction (Experimental): From a standardized preparation cannabis Cannabis FM2 (THC) (~ 6%) and (CBD) (~ 8%) ,cannabis decoction will be prepared at the moment by putting female inflorescences in cold water brought to a boil, boiling for 15 minutes and using 500 mg of medicinal cannabis for 500 ml of water.
  Interventions: Drug: Cannabis decoction
- Oral formulation: Cannabis oil (Experimental): From a standardized preparation cannabis Cannabis FM2 (THC) (~ 6%) and (CBD) (~ 8%), cannabis oil is prepared the day before the experimental session with 500 mg of female inflorescences in 5 ml of olive oil from the European Pharmacopoeia, heating in a water bath (approximately 98 ° C) for 120 minutes and cooling the oil samples. at room temperature.
  Interventions: Drug: Cannabis oil
- Vaporized formulation: Cannabis vaporized (Experimental): From a standardized preparation cannabis Cannabis FM2 (THC) (~ 6%) and (CBD) (~ 8%), 100 mg of Cannabis inflorescences of FM2 standardized cannabis were administered through Volcano vaporizer .
  Interventions: Drug: Vaporized cannabis

INTERVENTIONS:
Drug: Cannabis decoction — A single 100 mL dose of cannabis decoction is administered containing 1.8 mg THC and 2.7 mg CBD.
  Other Names: Cannabis tea
  Arms: Oral formulation: Cannabis decoction
Drug: Cannabis oil — A single administration of 15 drops (045 mL) of cannabis oil containing 1.8 mg THC and 3.8 mg CBD.
  Arms: Oral formulation: Cannabis oil
Drug: Vaporized cannabis — 100mg of vaporized cannabis is administered by Volcano vaporizer, wich containing 0.6-2 mg THC and 0.8-3 mg CBD
  Other Names: Inhaled cannabis
  Arms: Vaporized formulation: Cannabis vaporized

SUMMARY:
The purposes of the study are 1) to know the concentrations of Δ9-tetrahydrocannabinol (THC), cannabidiol (CBD) and other cannabinoids in blood, urine, oral fluid and sweat after the experimental administration of a standardized cannabis preparation orally (decoction and oil) and vaporized 2) to evaluate the pharmacological acute effects and tolerability

DETAILED DESCRIPTION:
Medical cannabis" encompasses the use of cannabis and cannabinoids for therapeutic purposes. Includes drugs approved by regulatory agencies and pharmaceutical products. Recently, many countries have authorized the use of cannabis flower cups with a standardized amount of Δ9-tetrahydrocannabinol (THC), cannabidiol (CBD) and their acidic precursors (Δ-9-tetrahydrocannabinolic acid A [THCA] and cannabidiol acid [ CBDA]) for the treatment of different diseases. In Italy since January 2017 there has been for sale a standardized cannabis preparation produced by the Military Pharmaceutical Institute of Florence. This medicinal variety of cannabis sativa, known as FM2 has a variable THC and CBD percentage of between 5-8% and 7-12% respectively. To date, there are no studies on the pharmacokinetics of THC, CBD and other minor cannabinoids in conventional and unconventional biological matrices after oral administration of cannabis tea, cannabis oil and vaporized with the same medicinal preparation (FM2). The main objective is to know the concentrations of THC, CBD and metabolites, and other cannabinoids in blood, urine, oral fluid and sweat after the experimental administration of a standardized cannabis preparation orally (two formulations: cannabis tea and cannabis oil) and vaporized. In addition, the acute pharmacological effects and tolerability will be evaluated. Healthy recreational cannabis users with experience in oral use of cannabis will participate

ELIGIBILITY:
Inclusion Criteria:

* Understanding and accepting the study procedures and signing the informed consent.
* Male and females healthy volunteers (18-45 years old.
* History and physical examination showing no organic or psychiatric disorders.
* The EKG and the blood chemistry and hematology at inclusion must be within the limits of normality. Minor or specific variations of the limits of normality are admitted if, in the opinion of the Principal Investigator, taking into account the state of science, they do not have clinical significance, do not pose a risk to the subjects and do not interfere with the evaluation of the product. These variations and their non-relevance will be specifically justified in writing.
* Body weight between 50-90 kilograms. Lower or higher weights are allowed, in the opinion of the Principal Investigator or the collaborators designated by him and that do not pose a risk to the subjects and do not interfere with the objectives of the study.
* BMI between 19-27 kg / m². Lower or higher BMIs are admitted, which in the opinion of the Principal Investigator or the collaborators designated by him that do not pose a risk to the subjects and do not interfere with the objectives of the study.
* Women with a menstrual cycle that lasts between 26-32 days and is regular.
* Subjects with social or recreational consumption of cannabis in the last 12 months and consumption of oral cannabis at least once in their life (eg cake, cookies, oils, infusion…).

Exclusion Criteria:

* Not meeting the inclusion criteria.
* History or clinical evidence of gastrointestinal, liver, kidney or other disorders that may involve an alteration in the absorption, distribution, metabolism or excretion of the drug, or that are suggestive of gastrointestinal irritation by drugs.
* Current or previous history of Diagnostic and Statistical Manual of Mental Disorders V (DSM-V) substance use disorder (except nicotine and mild cannabis use disorder or DSM-IV for substance use disorder or abuse).
* Having donated blood in the previous 8 weeks, or having participated in clinical trials with drugs or nutraceuticals in the previous 12 weeks, except for having previously participated in this same study, in which a 3-week washout period is sufficient.
* Having suffered any organic disease or major surgery in the three months prior to the start of the study.
* Subjects who are intolerant or have had serious adverse reactions to cannabis.
* Having taken medication regularly in the month prior to the study sessions, with the exception of vitamins, herbal remedies or dietary supplements that, in the opinion of the Principal Investigator or the collaborators designated by him, do not pose a risk to the subjects and do not interfere with the objectives of the study. Treatment with single doses of symptomatic medication in the week prior to the study sessions will not be grounds for exclusion if it is assumed that it has been completely eliminated on the day of the experimental session.
* Smokers of more than 15 cigarettes a day.
* Subjects who are uncapable of understanding the nature of the trial and the procedures they are required to follow.
* Subjects with positive serology for hepatitis B, C or HIV.
* Women who are pregnant or breastfeeding, or who use hormonal contraceptives or do not use reliable contraceptive measures during the study (such as abstinence, intrauterine devices, barrier methods or with a vasectomized partner).
* Women with amenorrhea or severe premenstrual syndrome.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Maximum serum concentration (Cmax) of THC | From baseline to 24 hours after decoction, oil or vaporized cannabis administration.
  Calculation of maximum concentration (ng/mL) in samples collected from 15 min prior to administration (time zero) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after oral cannabis formulation ( decoction or oil). In the case of vaporized cannabis, serum samples are collected 15 minutes before, at time zero (administration), and at 10, 20, 40, 1, 1.5,2,3,4,6,8 and 24 hours.
Maximum serum concentration (Cmax) of THCA | From baseline to 24 hours after decoction, oil or vaporized cannabis administration.
  Calculation of maximum concentration (ng/mL) in samples collected from 15 min prior to administration (time zero) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after oral cannabis formulation ( decoction or oil). In the case of vaporized cannabis, serum samples are collected 15 minutes before, at time zero (administration), and at 10, 20, 40, 1, 1.5,2,3,4,6,8 and 24 hours.
Maximum serum concentration (Cmax) of CBD | From baseline to 24 hours after decoction, oil or vaporized cannabis administration.
  Calculation of maximum concentration (ng/mL) in samples collected from 15 min prior to administration (time zero) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after oral cannabis formulation ( decoction or oil). In the case of vaporized cannabis, serum samples are collected 15 minutes before, at time zero (administration), and at 10, 20, 40, 1, 1.5,2,3,4,6,8 and 24 hours.
Maximum serum concentration (Cmax) of CBDA | From baseline to 24 hours after decoction, oil or vaporized cannabis administration.
  Calculation of maximum concentration (ng/mL) in samples collected from 15 min prior to administration (time zero) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after oral cannabis formulation ( decoction or oil). In the case of vaporized cannabis, serum samples are collected 15 minutes before, at time zero (administration), and at 10, 20, 40, 1, 1.5,2,3,4,6,8 and 24 hours.
Time to reach maximum serum concentration (Tmax) of THC | From baseline to 24 hours after decoction, oil or vaporized cannabis administration.
  Time to reach maximun concentration after decoction, oil or vaporized cannabis formulations.
Time to reach maximum serum concentration (Tmax) of THCA | From baseline to 24 hours after decoction, oil or vaporized cannabis administration.
  Time to reach maximun concentration after decoction, oil or vaporized cannabis formulations.
Time to reach maximum serum concentration (Tmax) of THC metabolites | From baseline to 24 hours after decoction, oil or vaporized cannabis administration.
  Time to reach maximun concentration after decoction, oil or vaporized cannabis formulations.
Time to reach maximum serum concentration (Tmax) of CBD | From baseline to 24 hours after decoction, oil or vaporized cannabis administration.
  Time to reach maximun concentration after decoction, oil or vaporized cannabis formulations.
Time to reach maximum serum concentration (Tmax) of CBDA | From baseline to 24 hours after decoction, oil or vaporized cannabis administration.
  Time to reach maximun concentration after decoction, oil or vaporized cannabis formulations.
Area under the concentration-time curve (AUC 0-24 h) of THC in serum concentrations | From baseline to 24 hours after administration ( decoction, oil or vaporized cannabis )
  Calculation of AUC with samples collected from 15 min prior to administration (time zero) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after oral cannabis formulation ( decoction or oil). In the case of vaporized cannabis, serum samples are collected 15 minutes before, at time zero (administration), and at 10, 20, 40, 1, 1.5,2,3,4,6,8 and 24 hours.
Area under the concentration-time curve (AUC 0-24 h) of THCA in serum concentrations | From baseline to 24 hours after administration ( decoction, oil or vaporized cannabis )
  Calculation of AUC with samples collected from 15 min prior to administration (time zero) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after oral cannabis formulation ( decoction or oil). In the case of vaporized cannabis, serum samples are collected 15 minutes before, at time zero (administration), and at 10, 20, 40, 1, 1.5,2,3,4,6,8 and 24 hours.
Area under the concentration-time curve (AUC 0-24 h) of CBD in serum concentrations | From baseline to 24 hours after administration ( decoction, oil or vaporized cannabis )
  Calculation of AUC with samples collected from 15 min prior to administration (time zero) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after oral cannabis formulation ( decoction or oil). In the case of vaporized cannabis, serum samples are collected 15 minutes before, at time zero (administration), and at 10, 20, 40, 1, 1.5,2,3,4,6,8 and 24 hours.
Area under the concentration-time curve (AUC 0-24 h) of CBDA in serum concentrations | From baseline to 24 hours after administration ( decoction, oil or vaporized cannabis )
  Calculation of AUC with samples collected from 15 min prior to administration (time zero) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after oral cannabis formulation ( decoction or oil). In the case of vaporized cannabis, serum samples are collected 15 minutes before, at time zero (administration), and at 10, 20, 40, 1, 1.5,2,3,4,6,8 and 24 hours.

SECONDARY OUTCOMES:
Maximum oral fluid concentration (Cmax) of THC | From baseline to 24 hours after decoction, oil or vaporized cannabis administration
  Calculation of maximum concentration (ng/mL) oral fluid samples collected with a Salivette device at the same time points as serum. Ora liquid is collected 15 min before administration (time zero), at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after the oral formulation of cannabis (decoction or oil) and in the case of vaporized cannabis at 15 minutes before zero time (administration), at 10, 20, 40, 1, 1.5,2,3,4,6,8 and 24 hours
Maximum oral fluid concentration (Cmax) of THCA | From baseline to 24 hours after decoction, oil or vaporized cannabis administration
  Calculation of maximum concentration (ng/mL) oral fluid samples collected with a Salivette device at the same time points as serum. Ora liquid is collected 15 min before administration (time zero), at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after the oral formulation of cannabis (decoction or oil) and in the case of vaporized cannabis at 15 minutes before zero time (administration), at 10, 20, 40, 1, 1.5,2,3,4,6,8 and 24 hours
Maximum oral fluid concentration (Cmax) of CBD | From baseline to 24 hours after decoction, oil or vaporized cannabis administration
  Calculation of maximum concentration (ng/mL) oral fluid samples collected with a Salivette device at the same time points as serum. Ora liquid is collected 15 min before administration (time zero), at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after the oral formulation of cannabis (decoction or oil) and in the case of vaporized cannabis at 15 minutes before zero time (administration), at 10, 20, 40, 1, 1.5,2,3,4,6,8 and 24 hours
Maximum oral fluid concentration (Cmax) of CBDA | From baseline to 24 hours after decoction, oil or vaporized cannabis administration
  Calculation of maximum concentration (ng/mL) oral fluid samples collected with a Salivette device at the same time points as serum. Ora liquid is collected 15 min before administration (time zero), at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after the oral formulation of cannabis (decoction or oil) and in the case of vaporized cannabis at 15 minutes before zero time (administration), at 10, 20, 40, 1, 1.5,2,3,4,6,8 and 24 hours
Time to reach maximum oral fluid concentration (Tmax) of THC | From baseline to 24 hours after decoction, oil or vaporized cannabis administration
  Time to reach maximun concentration after decoction, oil or vaporized cannabis formulations
Time to reach maximum oral fluid concentration (Tmax) of THCA | From baseline to 24 hours after decoction, oil or vaporized cannabis administration
  Time to reach maximun concentration after decoction, oil or vaporized cannabis formulations
Time to reach maximum oral fluid concentration (Tmax) of CBD | From baseline to 24 hours after decoction, oil or vaporized cannabis administration
  Time to reach maximun concentration after decoction, oil or vaporized cannabis formulations
Time to reach maximum oral fluid concentration (Tmax) of CBDA | From baseline to 24 hours after decoction, oil or vaporized cannabis administration
  Time to reach maximun concentration after decoction, oil or vaporized cannabis formulations
Area under the concentration-time curve (AUC 0-24h) of THC oral fluid concentrations | From baseline to 24 hours after decoction, oil or vaporized cannabis administration
  Calculation of AUC with samples collected from 15 min prior to administration (time zero) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after oral cannabis formulation ( decoction or oil). In the case of vaporized cannabis, serum samples are collected 15 minutes before, at time zero (administration), and at 10, 20, 40, 1, 1.5,2,3,4,6,8 hours
Area under the concentration-time curve (AUC 0-24h) of THCA oral fluid concentrations | From baseline to 24 hours after decoction, oil or vaporized cannabis administration
  Calculation of AUC with samples collected from 15 min prior to administration (time zero) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after oral cannabis formulation ( decoction or oil). In the case of vaporized cannabis, serum samples are collected 15 minutes before, at time zero (administration), and at 10, 20, 40, 1, 1.5,2,3,4,6,8 hours
Area under the concentration-time curve (AUC 0-24h) of CBD oral fluid concentrations | From baseline to 24 hours after decoction, oil or vaporized cannabis administration
  Calculation of AUC with samples collected from 15 min prior to administration (time zero) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after oral cannabis formulation ( decoction or oil). In the case of vaporized cannabis, serum samples are collected 15 minutes before, at time zero (administration), and at 10, 20, 40, 1, 1.5,2,3,4,6,8 hours
Area under the concentration-time curve (AUC 0-24h) of CBDA oral fluid concentrations | From baseline to 24 hours after decoction, oil or vaporized cannabis administration
  Calculation of AUC with samples collected from 15 min prior to administration (time zero) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours after oral cannabis formulation ( decoction or oil). In the case of vaporized cannabis, serum samples are collected 15 minutes before, at time zero (administration), and at 10, 20, 40, 1, 1.5,2,3,4,6,8 hours
Total amount cannabis metabolites (THC-carboxy and THC-glucoronides, excreted in 24 h urine samples. | From baseline to 24 hours after decoction, oil or vaporized cannabis administration
  Urine was collected 15 minutes before administration (time zero) and then between 0-2 h, 2-4 h, 6 h-8 h, 8-10 h, and 10-24 h after administration of oral and vaporized formulations.
Total concentration of THC present in sweat after oral and vaporized cannabis administration. | From baseline to 24 hours after decoction, oil or vaporized cannabis administration
  Concentration in ng/patch. Samples were collected with dermal patches (5 x 5 cm areas) applied to the back and removed at different intervals such as: 0-2 h, 2-4 h, 4-6 h, 6-8 h, 8-10 h, 10-12 h and 12-24 h
Total concentration of CBD present in sweat after oral and vaporized cannabis administration. | From baseline to 24 hours after decoction, oil or vaporized cannabis administration
  Concentration in ng/patch. Samples were collected with dermal patches (5 x 5 cm areas) applied to the back and removed at different intervals such as: 0-2 h, 2-4 h, 4-6 h, 6-8 h, 8-10 h, 10-12 h and 12-24 h
Change in blood pressure: Emax (peak/maximum effects) in blood pressure | Differences from baseline to 24 hours
  Non-invasive systolic blood pressure (mmHg) and diastolic blood pressure (mmHg) were repeatedly recorded at baseline (45 and 15 min) prior to decoction or oil administration, and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 h after administration. In case o vaporized cannabis were recorded at baseline (45 and 15 min) before and 10, 20, 40 min and 1, 1.5, 2, 3, 4, 6, 8, and 24 h after administration.
  Blood pressure measured in mmHg.
  .
Change in Heart rate: Emax (peak/maximum effects) in Heart rate | Differences from baseline to 24 hours
  Heart rate were repeatedly recorded at baseline (45 and 15 min) prior to decoction or oil administration, and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 h after administration. In case of vaporized cannabis were recorded at baseline (45 and 15 min) before and 10, 20, 40 min and 1, 1.5, 2, 3, 4, 6, 8, and 24 h after administration .
  Heart rate measured in beats per minute (bpm).
Change in oral temperature: Emax (peak/maximum effects) in oral temperature | Differences from baseline to 24 hours
  Oral temperature were repeatedly recorded at baseline (45 and 15 min) prior to decoction or oil administration, and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 h after administration. In case o vaporized cannabis were recorded at baseline (45 and 15 min) before and 10, 20, 40 min and 1, 1.5, 2, 3, 4, 6, 8, and 24 h after administration .
  Oral temperature measured in Celsius degrees (ºC).
Change in Intensity of effects: Emax (peak/maximum effects) in Intensity of effects | Differences from baseline to 24 hours
  Intensity of effects will be measured using a visual analog scale (0-100 mm) at baseline and 0.30, 1, 1.30, 2, 3, 4, 6,8, 10 and 24 h after oral cannabis administration, and at baseline ,10, 20, 40 min and 1, 1.5, 2, 3, 4, 6, 8, and 24 h after vaporized cannabis administration.
  Higher mm means more intensity of effects.
Change in High feeling: Emax (peak/maximum effects) in High feeling | Differences from baseline to 24 hours
  High will be measured using a visual analog scale 0-100 mm) at baseline and 0.30, 1, 1.30, 2, 3, 4, 6,8, 10 and 24 h after oral cannabis administration , and at baseline ,10, 20, 40 min and 1, 1.5, 2, 3, 4, 6, 8, and 24 h after vaporized cannabis administration.
  Higher mm means more high feeling.
Change in Hunger: Emax (peak/maximum effects) in Hunger | Differences from baseline to 24 hours
  Hunger will be measured using a visual analog scale (0-100 mm) at baseline and 0.30, 1, 1.30, 2, 3, 4, 6,8, 10 and 24 h after oral cannabis administration , and at baseline ,10, 20, 40 min and 1, 1.5, 2, 3, 4, 6, 8, and 24 h after vaporized cannabis administration.
  Higher mm means more hunger.
Change in Drowsines: Emax (peak/maximum effects) in Drowsiness | Differences from baseline to 24 hours
  Drowsiness will be measured using a visual analog scale (0-100 mm) at baseline and 0.30, 1, 1.30, 2, 3, 4, 6,8, 10 and 24 h after oral cannabis administration , and at baseline ,10, 20, 40 min and 1, 1.5, 2, 3, 4, 6, 8, and 24 h after vaporized cannabis administration.
  Higher mm means more drowsiness.
Change in global drug effects: Emax (peak/maximum effects) in global drug effects | Differences from baseline to 24 hours
  Global drug effects will be measured using the short form (49 items) of the Addiction Research Center Inventory (ARCI) . This is a true/false response questionnaire with 49 items. The global results include five subscales (sedation, euphoria, dysphoria, intellectual efficiency and amphetamine-like effects.
  It is administered at baseline and 0.30, 1, 1.30, 2, 3, 4, 6,8, 10 and 24 h after oral cannabis administration , and at baseline, 20, 40 min and 1, 1.5, 2, 3, 4, 6, 8, and 24 h after vaporized cannabis administration.
  Scores range usually from a total of 12 to 57 points. More points mean more effects.

CONTACTS AND LOCATIONS:
Overall Officials: Magi Farré, MD, PhD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Busardo FP, Perez-Acevedo AP, Pacifici R, Mannocchi G, Gottardi M, Papaseit E, Perez-Mana C, Martin S, Poyatos L, Pichini S, Farre M. Disposition of Phytocannabinoids, Their Acidic Precursors and Their Metabolites in Biological Matrices of Healthy Individuals Treated with Vaporized Medical Cannabis. Pharmaceuticals (Basel). 2021 Jan 13;14(1):59. doi: 10.3390/ph14010059. PMID 33451073
- [Result] Perez-Acevedo AP, Busardo FP, Pacifici R, Mannocchi G, Gottardi M, Poyatos L, Papaseit E, Perez-Mana C, Martin S, Di Trana A, Pichini S, Farre M. Disposition of Cannabidiol Metabolites in Serum and Urine from Healthy Individuals Treated with Pharmaceutical Preparations of Medical Cannabis. Pharmaceuticals (Basel). 2020 Dec 12;13(12):459. doi: 10.3390/ph13120459. PMID 33322849
- [Result] Pichini S, Malaca S, Gottardi M, Perez-Acevedo AP, Papaseit E, Perez-Mana C, Farre M, Pacifici R, Tagliabracci A, Mannocchi G, Busardo FP. UHPLC-MS/MS analysis of cannabidiol metabolites in serum and urine samples. Application to an individual treated with medical cannabis. Talanta. 2021 Feb 1;223(Pt 2):121772. doi: 10.1016/j.talanta.2020.121772. Epub 2020 Oct 14. PMID 33298281
- [Result] Perez-Acevedo AP, Pacifici R, Mannocchi G, Gottardi M, Poyatos L, Papaseit E, Perez-Mana C, Martin S, Busardo FP, Pichini S, Farre M. Disposition of cannabinoids and their metabolites in serum, oral fluid, sweat patch and urine from healthy individuals treated with pharmaceutical preparations of medical cannabis. Phytother Res. 2021 Mar;35(3):1646-1657. doi: 10.1002/ptr.6931. Epub 2020 Nov 6. PMID 33155722